CLINICAL TRIAL: NCT02819453
Title: Corticosteroid Treatment for Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director of respiratory department, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20150101
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: corticosteroid; acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prior corticosteroid treatment: Patients diagnosed with acute respiratory distress syndrome(ARDS) by two clinicians on the first day of hospital admission (not receiving corticosteroids yet)
- after corticosteroid treatment: Patients diagnosed with acute respiratory distress syndrome(ARDS) after corticosteroids treatment

SUMMARY:
It is acknowledged that IL-18, as a product of the inflammasome, is involved in host defence against viral and bacterial stimuli by modulating the immune response. The aim of this study was to determine IL-18 levels in serum of patients with acute respiratory distress syndrome and to investigate whether corticosteroid attenuate its levels. In addition, to explore the effect of corticosteroid therapy on the prognosis of ARDS.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is caused by an inflammatory injury to the lung that is characterized clinically by acute hypoxemic respiratory failure. Pathologically complex changes in the lung are manifested by an early, exudative phase followed by proliferative and fibrotic phases. Persistent ARDS is characterized by ongoing inflammation, parenchymal-cell proliferation, and disordered deposition of collagen, all of which may be responsive to corticosteroid therapy. Systemic corticosteroids have been considered a potentially beneficial therapy. However, several studies have failed to provide convincing evidence to prove the efficacy of corticosteroids in decreasing the mortality of ARDS. For the secondary outcomes, such as oxygenation improvement and reduction of the duration of mechanical ventilation, have shown consistent findings in favor of corticosteroid therapy. However, the underlying mechanisms that account for the anti-inflammatory actions of corticosteroid in ARDS patients have not yet to be elucidated, and the activities do not appear to be controlled by a single mechanism. Interleukin-18 (IL-18), along with interleukin-1b (IL-1b), is produced by inflammasomes when activated by a number of pathogen, environmental or host-derived danger signals. Inflammasomes are innate immune regulatory protein complexes which seem to play a key role in the host immune response of patients with ARDS. The aim of this study is to determine the role of steroid on IL-18 levels in serum of patients with ARDS and its effect on prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent;
2. Aged 18-85 years;
3. Confirmed diagnosis of ARDS by Berlin criterion

Exclusion Criteria:

1. Active tuberculosis and disseminated fungal infection;
2. Chronic corticosteroid application
3. Patients with organ dysfunction, such as severe liver dysfunction, adrenal insufficiency, severe cardiopulmonary dysfunction;
4. Hypogammaglobulinemia or other autoimmune disease;
5. Acquired immunodeficiency syndrome;
6. Refuse to use corticosteroid;
7. Pregnant or nursing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients diagnosed with acute respiratory distress syndrome (ARDS) based on Berlin criterion by two clinicians
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
serum IL-18 level | three days
  the serum IL-18 level of ARDS patients detected by Human IL-18 ELISA kit prior and after corticosteroid treatment
arterial partial pressure of oxygen/ fraction of inspired oxygen (PaO2/FiO2) | three days
  arterial partial pressure of oxygen/ fraction of inspired oxygen (PaO2/FiO2) prior and after corticosteroid treatment
the acute physiology and chronic health evaluation (APACHE II) score | seven days
  the acute physiology and chronic health evaluation (APACHE II) score prior and after corticosteroid treatment. This score system on a scale range from 0 to 71 scores, the higher scores mean a worse outcome.
the ratio of Neutrophils/lymphocyte | three days
  the ratio of Neutrophils/lymphocyte prior and after corticosteroid treatment
45-day mortality after corticosteroid treatment | 45 days
  45-day mortality of ARDS patients after corticosteroid treatment

SECONDARY OUTCOMES:
factors associated with the mortality of ARDS patients | 45 days
  factors associated with the mortality of ARDS patients

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, PhD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital , Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Dolinay T, Kim YS, Howrylak J, Hunninghake GM, An CH, Fredenburgh L, Massaro AF, Rogers A, Gazourian L, Nakahira K, Haspel JA, Landazury R, Eppanapally S, Christie JD, Meyer NJ, Ware LB, Christiani DC, Ryter SW, Baron RM, Choi AM. Inflammasome-regulated cytokines are critical mediators of acute lung injury. Am J Respir Crit Care Med. 2012 Jun 1;185(11):1225-34. doi: 10.1164/rccm.201201-0003OC. Epub 2012 Mar 29. PMID 22461369
- [Derived] Yang JW, Jiang P, Wang WW, Wen ZM, Mao B, Lu HW, Zhang L, Song YL, Xu JF. The Controversy About the Effects of Different Doses of Corticosteroid Treatment on Clinical Outcomes for Acute Respiratory Distress Syndrome Patients: An Observational Study. Front Pharmacol. 2021 Jul 29;12:722537. doi: 10.3389/fphar.2021.722537. eCollection 2021. PMID 34393800
- [Derived] Sweeney RM, McAuley DF. Prolonged glucocorticoid treatment in acute respiratory distress syndrome - Authors' reply. Lancet. 2017 Apr 15;389(10078):1516-1517. doi: 10.1016/S0140-6736(17)30953-4. No abstract available. PMID 28422025